CLINICAL TRIAL: NCT02595528
Title: A Phase 2, Multicenter, Double-masked, Randomized, Vehicle-Controlled, Study of the Concurrent Use of AGN-190584 and AGN-199201 in Patients With Presbyopia
Brief Title: A Study of the Concurrent Use of AGN-190584 and AGN-199201 in Participants With Presbyopia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 199201-009
Record Dates: First submitted 2015-11-02; First posted 2015-11-03 (Estimated); Results first posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-11

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AGN-199201 and AGN-190584 Vehicle (Experimental): Participants will receive 5 different treatments as per protocol for 2 days each. Treatment 1: nondominant eye--1 drop AGN-199201 vehicle followed by 1 drop AGN-190584 vehicle, dominant eye--2 drops AGN-190584 vehicle; Treatment 2: nondominant eye--1 drop AGN-199201 Dose A followed by 1 drop AGN-190584 vehicle, dominant eye--2 drops AGN-190584 vehicle; Treatment 3: nondominant eye--1 drop AGN-199201 Dose B followed by 1 drop AGN-190584 vehicle, dominant eye--2 drops AGN-190584 vehicle; Treatment 4: nondominant eye--1 drop AGN-199201 Dose C followed by 1 drop AGN-190584 vehicle, dominant eye--2 drops AGN-190584 vehicle; Treatment 5: nondominant eye--1 drop fixed combination of AGN-199201 and AGN-190584 followed by 1 drop AGN-190584 vehicle, dominant eye--2 drops AGN-190584 vehicle.
  Interventions: Drug: AGN-199201 ophthalmic solution; Drug: AGN-190584 ophthalmic solution; Drug: AGN-190584 vehicle; Drug: AGN-199201 + AGN-190584 Combination; Drug: AGN-199201 vehicle
- AGN-199201 and AGN-190584 Dose A (Experimental): Participants will receive 5 different treatments as per protocol for 2 days each. Treatment 1: nondominant eye--1 drop AGN-199201 vehicle followed by 1 drop AGN-190584 Dose A, dominant eye--2 drops AGN-190584 vehicle; Treatment 2: nondominant eye--1 drop AGN-199201 Dose A followed by 1 drop AGN-190584 Dose A, dominant eye--2 drops AGN-190584 vehicle; Treatment 3: nondominant eye--1 drop AGN-199201 Dose B followed by 1 drop AGN-190584 Dose A, dominant eye--2 drops AGN-190584 vehicle; Treatment 4: nondominant eye--1 drop AGN-199201 Dose C followed by 1 drop AGN-190584 Dose A, dominant eye--2 drops AGN-190584 vehicle; Treatment 5: nondominant eye--1 drop fixed combination of AGN-199201 and AGN-190584 followed by 1 drop AGN-190584 vehicle, dominant eye--2 drops AGN-190584 vehicle.
  Interventions: Drug: AGN-199201 ophthalmic solution; Drug: AGN-190584 ophthalmic solution; Drug: AGN-190584 vehicle; Drug: AGN-199201 + AGN-190584 Combination; Drug: AGN-199201 vehicle
- AGN-199201 and AGN-190584 Dose B (Experimental): Participants will receive 5 different treatments as per protocol for 2 days each. Treatment 1: nondominant eye--1 drop AGN-199201 vehicle followed by 1 drop AGN-190584 Dose B, dominant eye--2 drops AGN-190584 vehicle; Treatment 2: nondominant eye--1 drop AGN-199201 Dose A followed by 1 drop AGN-190584 Dose B, dominant eye--2 drops AGN-190584 vehicle; Treatment 3: nondominant eye--1 drop AGN-199201 Dose B followed by 1 drop AGN-190584 Dose B, dominant eye--2 drops AGN-190584 vehicle; Treatment 4: nondominant eye--1 drop AGN-199201 Dose C followed by 1 drop AGN-190584 Dose B, dominant eye--2 drops AGN-190584 vehicle; Treatment 5: nondominant eye--1 drop fixed combination of AGN-199201 and AGN-190584 followed by 1 drop AGN-190584 vehicle, dominant eye--2 drops AGN-190584 vehicle.
  Interventions: Drug: AGN-199201 ophthalmic solution; Drug: AGN-190584 ophthalmic solution; Drug: AGN-190584 vehicle; Drug: AGN-199201 + AGN-190584 Combination; Drug: AGN-199201 vehicle
- AGN-199201 and AGN-190584 Dose C (Experimental): Participants will receive 5 different treatments as per protocol for 2 days each. Treatment 1: nondominant eye--1 drop AGN-199201 vehicle followed by 1 drop AGN-190584 Dose C, dominant eye--2 drops AGN-190584 vehicle; Treatment 2: nondominant eye--1 drop AGN-199201 Dose A followed by 1 drop AGN-190584 Dose C, dominant eye--2 drops AGN-190584 vehicle; Treatment 3: nondominant eye--1 drop AGN-199201 Dose B followed by 1 drop AGN-190584 Dose C, dominant eye--2 drops AGN-190584 vehicle; Treatment 4: nondominant eye--1 drop AGN-199201 Dose C followed by 1 drop AGN-190584 Dose C, dominant eye--2 drops AGN-190584 vehicle; Treatment 5: nondominant eye--1 drop fixed combination of AGN-199201 and AGN-190584 followed by 1 drop AGN-190584 vehicle, dominant eye--2 drops AGN-190584 vehicle.
  Interventions: Drug: AGN-199201 ophthalmic solution; Drug: AGN-190584 ophthalmic solution; Drug: AGN-190584 vehicle; Drug: AGN-199201 + AGN-190584 Combination; Drug: AGN-199201 vehicle

INTERVENTIONS:
Drug: AGN-199201 ophthalmic solution — 1 drop of AGN-199201 ophthalmic solution Doses A, B, C in the eye.
Drug: AGN-190584 ophthalmic solution — 1 drop AGN-190584 ophthalmic solution doses A, B and C in the eye.
Drug: AGN-190584 vehicle — Vehicle to AGN-190584
Drug: AGN-199201 + AGN-190584 Combination — 1 drop AGN-199201 and AGN-190584 fixed combination ophthalmic solution in the eye.
Drug: AGN-199201 vehicle — Vehicle to AGN-199201

SUMMARY:
This study will identify the optimum concentrations of AGN-199201 and AGN-190584 when dosed in combination once a day for the improvement of uncorrected near visual acuity in participants with presbyopia (inability to focus on items close-up).

ELIGIBILITY:
Inclusion Criteria:

-Normal vision at distance, either natural or post corneal laser refractive surgery, with presbyopia in each eye and complaints of poor near vision that impacts activities of daily living.

Exclusion Criteria:

* Use of any topical ophthalmic medications, including artificial tears other than the study medications during the study
* Corneal abnormalities in either eye that interfere with visual acuity
* History of cataract surgery, phakic intraocular lens surgery, corneal inlay surgery or any intraocular surgery
* Diagnosis of glaucoma or ocular hypertension.

Ages: 40 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 163 (Actual)
Dates: Start 2016-04-29 (Actual); Primary Completion 2017-10-18 (Actual); Study Completion 2017-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haixia Liu, Study Director — Allergan
Locations (20):
- United States (20):
  - Sall Research Medical Center, Artesia, California
  - Milton M. Hom, OD, FAAO, Azusa, California
  - WCCT Global, LLC, Costa Mesa, California
  - The Eye Research Foundation, Newport Beach, California
  - North Bay Eye Associates, Inc., Petaluma, California
  - Martel Eye Medical Group, Rancho Cordova, California
  - West Coast Eye Care, San Diego, California
  - Corneal Consultants of Colorado, P.C., Littleton, Colorado
  - Mid Florida Eye Center, Mt. Dora, Florida
  - Clayton Eye Center, Morrow, Georgia
  - Price Vision Group, Indianapolis, Indiana
  - Specialized Eye Care, Baltimore, Maryland
  - Comprehensive Eye Care, Ltd, Washington, Missouri
  - Cleveland Eye Clinic, Brecksville, Ohio
  - Scott & Christie and Associates, PC, Cranberry Township, Pennsylvania
  - Total Eye Care, PA, Memphis, Tennessee
  - Cataract and Glaucoma Center, El Paso, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Hoopes Durrie Rivera Research, LLC, Draper, Utah
  - The Eye Centers of Racine & Kenosha, Kenosha, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomization and treatment assignment were based on a randomization scheme prepared by Allergan Biostatistics prior to the start of the study.
Groups:
- AGN-190584 Vehicle and AGN-199201: Participants will receive 5 different treatments as per protocol for 2 days each. Treatment 1: nondominant eye--1 drop AGN-199201 vehicle followed by 1 drop AGN-190584 vehicle, dominant eye--2 drops AGN-190584 vehicle; Treatment 2: nondominant eye--1 drop AGN-199201 Lower Dose followed by 1 drop AGN-190584 vehicle, dominant eye--2 drops AGN-190584 vehicle; Treatment 3: nondominant eye--1 drop AGN-199201 Medium Dose followed by 1 drop AGN-190584 vehicle, dominant eye--2 drops AGN-190584 vehicle; Treatment 4: nondominant eye--1 drop AGN-199201 Higher Dose followed by 1 drop AGN-190584 vehicle, dominant eye--2 drops AGN-190584 vehicle; Treatment 5: nondominant eye--1 drop fixed combination of AGN-199201 and AGN-190584 followed by 1 drop AGN-190584 vehicle, dominant eye--2 drops AGN-190584 vehicle.
- AGN-190584 Lower Dose and AGN-199201: Participants will receive 5 different treatments as per protocol for 2 days each. Treatment 1: nondominant eye--1 drop AGN-199201 vehicle followed by 1 drop AGN-190584 Lower Dose, dominant eye--2 drops AGN-190584 vehicle; Treatment 2: nondominant eye--1 drop AGN-199201 Lower Dose followed by 1 drop AGN-190584 Lower Dose, dominant eye--2 drops AGN-190584 vehicle; Treatment 3: nondominant eye--1 drop AGN-199201 Medium Dose followed by 1 drop AGN-190584 Lower Dose, dominant eye--2 drops AGN-190584 vehicle; Treatment 4: nondominant eye--1 drop AGN-199201 Higher Dose followed by 1 drop AGN-190584 Lower Dose, dominant eye--2 drops AGN-190584 vehicle; Treatment 5: nondominant eye--1 drop fixed combination of AGN-199201 and AGN-190584 followed by 1 drop AGN-190584 vehicle, dominant eye--2 drops AGN-190584 vehicle.
- AGN-190584 Medium Dose and AGN-199201: Participants will receive 5 different treatments as per protocol for 2 days each. Treatment 1: nondominant eye--1 drop AGN-199201 vehicle followed by 1 drop AGN-190584 Medium Dose, dominant eye--2 drops AGN-190584 vehicle; Treatment 2: nondominant eye--1 drop AGN-199201 Lower Dose followed by 1 drop AGN-190584 Medium Dose, dominant eye--2 drops AGN-190584 vehicle; Treatment 3: nondominant eye--1 drop AGN-199201 Medium Dose followed by 1 drop AGN-190584 Medium Dose, dominant eye--2 drops AGN-190584 vehicle; Treatment 4: nondominant eye--1 drop AGN-199201 Higher Dose followed by 1 drop AGN-190584 Medium Dose, dominant eye--2 drops AGN-190584 vehicle; Treatment 5: nondominant eye--1 drop fixed combination of AGN-199201 and AGN-190584 followed by 1 drop AGN-190584 vehicle, dominant eye--2 drops AGN-190584 vehicle.
- AGN-190584 Higher Dose and AGN-199201: Participants will receive 5 different treatments as per protocol for 2 days each. Treatment 1: nondominant eye--1 drop AGN-199201 vehicle followed by 1 drop AGN-190584 Higher Dose, dominant eye--2 drops AGN-190584 vehicle; Treatment 2: nondominant eye--1 drop AGN-199201 Lower Dose followed by 1 drop AGN-190584 Higher Dose, dominant eye--2 drops AGN-190584 vehicle; Treatment 3: nondominant eye--1 drop AGN-199201 Medium Dose followed by 1 drop AGN-190584 Higher Dose, dominant eye--2 drops AGN-190584 vehicle; Treatment 4: nondominant eye--1 drop AGN-199201 Higher Dose followed by 1 drop AGN-190584 Higher Dose, dominant eye--2 drops AGN-190584 vehicle; Treatment 5: nondominant eye--1 drop fixed combination of AGN-199201 and AGN-190584 followed by 1 drop AGN-190584 vehicle, dominant eye--2 drops AGN-190584 vehicle.
Period: Overall Study
Arm/Group | AGN-190584 Vehicle and AGN-199201 | AGN-190584 Lower Dose and AGN-199201 | AGN-190584 Medium Dose and AGN-199201 | AGN-190584 Higher Dose and AGN-199201
Started | 41 | 40 | 42 | 40
Completed | 39 | 37 | 41 | 36
Not Completed | 2 | 3 | 1 | 4
Not completed — Withdrawal by Subject | 1 | 2 | 1 | 3
Not completed — Lost to Follow-up | 1 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population: all subjects who received ≥ 1 administration of study treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | AGN-190584 Vehicle and AGN-199201 | AGN-190584 Lower Dose and AGN-199201 | AGN-190584 Medium Dose and AGN-199201 | AGN-190584 Higher Dose and AGN-199201 | Total
Number analyzed (Participants) | 41 | 39 | 42 | 39 | 161
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.6 (2.9) | 47.1 (2.7) | 46.8 (2.8) | 46.7 (2.3) | 46.8 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 27 | 29 | 24 | 112
  Male | 9 | 12 | 13 | 15 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 11 | 3 | 9 | 30
  Not Hispanic or Latino | 34 | 28 | 39 | 30 | 131
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 0 | 2
  Asian | 3 | 1 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 6 | 13 | 3 | 28
  White | 32 | 30 | 28 | 36 | 126
  More than one race | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Baseline UNVA severity [Count of Participants; unit: Participants] — Baseline UNVA measured visual acuity using Snellen Scores. Worse "severity" meant poorer visual acuity as measured by baseline UNVA (uncorrected near visual acuity). This graded measure was used to stratify participants into two groups: UNVA at baseline (≤ 20/80 and > 20/80).
  Participants
    ≤ 20/80 | 26 | 28 | 28 | 26 | 108
    > 20/80 | 15 | 11 | 14 | 13 | 53

OUTCOME MEASURES:

1. Primary Outcome: Weighted Average Change From Baseline in Mesopic, High Contrast Uncorrected Near Visual Acuity (UNVA) Letters
Description: UNVA is assessed without corrective lenses in the non-dominant eye. UNVA is measured using an eye chart and is reported as the number of lines read correctly. The lower the number of lines read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of lines read correctly means that vision has improved.
Time Frame: Baseline, Between hour 1 and hour 10 of each of the five 2-day dosing periods
Population: Modified Intent-to-Treat (mITT) population: all randomized patients who were randomized with a baseline and at least 1 post baseline assessment of mesopic, high contrast, UNVA.
Measure: Least Squares Mean (Standard Error); unit: letters correctly read
Groups:
- AGN-190584 Vehicle: Participants will receive 5 different treatments as per protocol for 2 days each. Treatment 1: nondominant eye--1 drop AGN-199201 vehicle followed by 1 drop AGN-190584 vehicle, dominant eye--2 drops AGN-190584 vehicle; Treatment 2: nondominant eye--1 drop AGN-199201 Lower Dose followed by 1 drop AGN-190584 vehicle, dominant eye--2 drops AGN-190584 vehicle; Treatment 3: nondominant eye--1 drop AGN-199201 Medium Dose followed by 1 drop AGN-190584 vehicle, dominant eye--2 drops AGN-190584 vehicle; Treatment 4: nondominant eye--1 drop AGN-199201 Higher Dose followed by 1 drop AGN-190584 vehicle, dominant eye--2 drops AGN-190584 vehicle; Treatment 5: nondominant eye--1 drop fixed combination of AGN-199201 and AGN-190584 followed by 1 drop AGN-190584 vehicle, dominant eye--2 drops AGN-190584 vehicle.
- AGN-190584 Lower Dose: Participants will receive 5 different treatments as per protocol for 2 days each. Treatment 1: nondominant eye--1 drop AGN-199201 vehicle followed by 1 drop AGN-190584 Lower Dose, dominant eye--2 drops AGN-190584 vehicle; Treatment 2: nondominant eye--1 drop AGN-199201 Lower Dose followed by 1 drop AGN-190584 Lower Dose, dominant eye--2 drops AGN-190584 vehicle; Treatment 3: nondominant eye--1 drop AGN-199201 Medium Dose followed by 1 drop AGN-190584 Lower Dose, dominant eye--2 drops AGN-190584 vehicle; Treatment 4: nondominant eye--1 drop AGN-199201 Higher Dose followed by 1 drop AGN-190584 Lower Dose, dominant eye--2 drops AGN-190584 vehicle; Treatment 5: nondominant eye--1 drop fixed combination of AGN-199201 and AGN-190584 followed by 1 drop AGN-190584 vehicle, dominant eye--2 drops AGN-190584 vehicle.
- AGN-190584 Medium Dose: Participants will receive 5 different treatments as per protocol for 2 days each. Treatment 1: nondominant eye--1 drop AGN-199201 vehicle followed by 1 drop AGN-190584 Medium Dose, dominant eye--2 drops AGN-190584 vehicle; Treatment 2: nondominant eye--1 drop AGN-199201 Lower Dose followed by 1 drop AGN-190584 Medium Dose, dominant eye--2 drops AGN-190584 vehicle; Treatment 3: nondominant eye--1 drop AGN-199201 Medium Dose followed by 1 drop AGN-190584 Medium Dose, dominant eye--2 drops AGN-190584 vehicle; Treatment 4: nondominant eye--1 drop AGN-199201 Higher Dose followed by 1 drop AGN-190584 Medium Dose, dominant eye--2 drops AGN-190584 vehicle; Treatment 5: nondominant eye--1 drop fixed combination of AGN-199201 and AGN-190584 followed by 1 drop AGN-190584 vehicle, dominant eye--2 drops AGN-190584 vehicle.
- AGN-190584 Higher Dose: Participants will receive 5 different treatments as per protocol for 2 days each. Treatment 1: nondominant eye--1 drop AGN-199201 vehicle followed by 1 drop AGN-190584 Higher Dose, dominant eye--2 drops AGN-190584 vehicle; Treatment 2: nondominant eye--1 drop AGN-199201 Lower Dose followed by 1 drop AGN-190584 Higher Dose, dominant eye--2 drops AGN-190584 vehicle; Treatment 3: nondominant eye--1 drop AGN-199201 Medium Dose followed by 1 drop AGN-190584 Higher Dose, dominant eye--2 drops AGN-190584 vehicle; Treatment 4: nondominant eye--1 drop AGN-199201 Higher Dose followed by 1 drop AGN-190584 Higher Dose, dominant eye--2 drops AGN-190584 vehicle; Treatment 5: nondominant eye--1 drop fixed combination of AGN-199201 and AGN-190584 followed by 1 drop AGN-190584 vehicle, dominant eye--2 drops AGN-190584 vehicle.
Arm/Group | AGN-190584 Vehicle | AGN-190584 Lower Dose | AGN-190584 Medium Dose | AGN-190584 Higher Dose
Number analyzed (Participants) | 40 | 37 | 42 | 38
letters correctly read
  AGN-199201 Vehicle: number analyzed (Participants) | 39 | 37 | 42 | 36
  AGN-199201 Vehicle | 1.12 (0.48) | 3.83 (0.37) | 5.26 (0.37) | 5.42 (0.50)
  AGN-199201 Lower Dose: number analyzed (Participants) | 38 | 35 | 41 | 36
  AGN-199201 Lower Dose | 1.24 (0.44) | 3.94 (0.34) | 5.37 (0.34) | 5.52 (0.46)
  AGN-199201 Medium Dose: number analyzed (Participants) | 39 | 35 | 41 | 35
  AGN-199201 Medium Dose | 1.47 (0.47) | 4.16 (0.39) | 5.56 (0.39) | 5.70 (0.48)
  AGN-199201 Higher Dose: number analyzed (Participants) | 39 | 35 | 41 | 37
  AGN-199201 Higher Dose | 1.34 (0.55) | 3.99 (0.41) | 5.36 (0.40) | 5.46 (0.56)
Statistical Analysis 1: Comparison: AGN-190584 Vehicle vs AGN-190584 Lower Dose vs AGN-190584 Medium Dose vs AGN-190584 Higher Dose; AGN-190584 Quadratic; Test type: Superiority; p = 0.0029, Mixed model for repeated measures; Least Squares (LS) = -2.5543
Statistical Analysis 2: Comparison: AGN-190584 Vehicle vs AGN-190584 Lower Dose vs AGN-190584 Medium Dose vs AGN-190584 Higher Dose; AGN-190584 Linear; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Least Squares (LS) = 6.6961
Statistical Analysis 3: Comparison: AGN-190584 Vehicle vs AGN-190584 Lower Dose vs AGN-190584 Medium Dose vs AGN-190584 Higher Dose; AGN-199201 Quadratic; Test type: Superiority; p = 0.4126, Mixed model for repeated measures; Least Squares (LS) = -69.890
Statistical Analysis 4: Comparison: AGN-190584 Vehicle vs AGN-190584 Lower Dose vs AGN-190584 Medium Dose vs AGN-190584 Higher Dose; AGN-199201 Linear; Test type: Superiority; p = 0.3752, Mixed model for repeated measures; Least Squares (LS) = 10.5017

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 112 days.
Description: Safety Population: all subjects who received ≥ 1 administration of study treatment.
Arm/Group | AGN-190584 Vehicle and AGN-199201 | AGN-190584 Lower Dose and AGN-199201 | AGN-190584 Medium Dose and AGN-199201 | AGN-190584 Higher Dose and AGN-199201
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/39 | 0/42 | 0/39
Serious Adverse Events (participants affected / at risk) | 1/41 | 1/39 | 0/42 | 1/39
Other Adverse Events (participants affected / at risk) | 9/41 | 9/39 | 16/42 | 17/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AGN-190584 Vehicle and AGN-199201 (N=41) | AGN-190584 Lower Dose and AGN-199201 (N=39) | AGN-190584 Medium Dose and AGN-199201 (N=42) | AGN-190584 Higher Dose and AGN-199201 (N=39)
Cervix carcinoma stage 0 (Investigations) | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Malignant melanoma (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AGN-190584 Vehicle and AGN-199201 (N=41) | AGN-190584 Lower Dose and AGN-199201 (N=39) | AGN-190584 Medium Dose and AGN-199201 (N=42) | AGN-190584 Higher Dose and AGN-199201 (N=39)
Instillation site pain (General disorders) | 3 | 0 | 1 | 3
Headache (Nervous system disorders) | 5 | 4 | 8 | 7
Lacrimation increased (Eye disorders) | 0 | 3 | 2 | 0
Foreign body sensation in eyes (Eye disorders) | 1 | 2 | 0 | 0
Punctate keratitis (Eye disorders) | 2 | 1 | 4 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 3 | 1
Visual impairment (Eye disorders) | 1 | 0 | 1 | 4
Visual acuity reduced (Eye disorders) | 0 | 0 | 1 | 2
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-11-09): https://cdn.clinicaltrials.gov/large-docs/28/NCT02595528/SAP_000.pdf
  • Study Protocol (2016-04-04): https://cdn.clinicaltrials.gov/large-docs/28/NCT02595528/Prot_001.pdf